CLINICAL TRIAL: NCT01023750
Title: Pretreatment Genotyping at APOA5 and GCKR Loci and Response to Fenofibrate Therapy
Brief Title: Predictors of Response to Fenofibrate
Acronym: PreFar
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Tufts University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: R21DK084560 (NIH)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2013-11

CONDITIONS: Hypertriglyceridemia; Insulin Resistance
Keywords: hypertriglyceridemia; Triglycerides; HDL; Insulin resistance
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance | interventions — Fenofibrate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fenofibrate
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — Participants will give a baseline blood sample and begin the 4 week course of fenofibrate. Patients will be given a 33-day dose of 145 mg of fenofibrate to be taken by mouth once a day. All doses of fenofibrate will be purchased in one batch, prepared at the pharmacy under supervision. A study nurse will collect each patient's 33-day dose of fenofibrate from the pharmacy and dispense to the study participants in the clinics. Patients will be given instructions on how to take the medication and given a 24-hr phone number to call in case of questions or need for additional care. Each patient will receive a phone call at least 2 times during the course of the trial to monitor the progress. Our co-investigators, who are also physicians will be available in case a study participant needs additional care. If not available, study participants will be able to reach the cardiologist or endocrinologist on call through an additional phone number we will provide.
  Other Names: Brand Name: TRICOR; NDC# 00074-6123-90

SUMMARY:
Fenofibrate is one of the best options for treating hypertriglyceridemia. In the majority of patients, fenofibrate lowers triglycerides (TG) by 24-55% and improves HDL- and LDL-cholesterol. However, the response to fenofibrate is highly variable and currently there are no screening tests to identify poor responders. Genetic and environmental factors may explain the high variability in response. Although exploratory in nature, this study is of clinical and public health importance because prediction of drug response among those with hypertriglyceridemia is clinically challenging and fenofibrate prescription costs are large ($90 to $130/patient/month); targeting the responsive patients at the outset will help improve treatment outcomes at a lower cost. If successful, the investigators will propose to conduct a large, randomized trial on the effect of pre-prescription genotyping on fenofibrate response.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or over dyslipidemic patients designated to receive fenofibrate by their attending physician.
* All patients will be seen at the UAB Diabetes and Endocrine Clinic or Cardiology Clinic.
* Women who are unable to have children because of surgery or other medical reason or are using an effective form of birth control before the study begins and agree to continue to use an effective form of birth control for 6 months after taking the study drug.

Exclusion Criteria:

* Under 19 and/or not a Dyslipidemic patient or dyslipidemic but with a medical condition (e.g., liver or kidney disease) that warrants contraindication of fenofibrate.
* Women who are pregnant, nursing and women who, unless they are unable to have children because of surgery or other medical reason, have not been using an effective form of birth control before the study begins and/or are unwilling to use an effective form of birth control for 6 months after taking the study drug will be excluded from the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are seen in the UAB Diabetes and Endocrine Clinic or Cardiology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in fasting triglyceride concentrations | 4 weeks

SECONDARY OUTCOMES:
Changes in lipids and markers of insulin resistance | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edmond K Kabagambe, DVM, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Lai CQ, Parnell LD, Lee YC, Zeng H, Smith CE, McKeown NM, Arnett DK, Ordovas JM. The impact of alcoholic drinks and dietary factors on epigenetic markers associated with triglyceride levels. Front Genet. 2023 Feb 15;14:1117778. doi: 10.3389/fgene.2023.1117778. eCollection 2023. PMID 36873949
- [Derived] Lai CQ, Parnell LD, Smith CE, Guo T, Sayols-Baixeras S, Aslibekyan S, Tiwari HK, Irvin MR, Bender C, Fei D, Hidalgo B, Hopkins PN, Absher DM, Province MA, Elosua R, Arnett DK, Ordovas JM. Carbohydrate and fat intake associated with risk of metabolic diseases through epigenetics of CPT1A. Am J Clin Nutr. 2020 Nov 11;112(5):1200-1211. doi: 10.1093/ajcn/nqaa233. PMID 32930325